CLINICAL TRIAL: NCT04114968
Title: Reducing the Burden of Cervical Cancer Among Older Women by Expanding the Screening Age and Offering HPV Self-sampling
Brief Title: Offering Cervical Cancer Screening to Older Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 2702
Record Dates: First submitted 2019-09-20; First posted 2019-10-03 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Uterine Cervical Neoplasm; Uterine Neoplasm; Uterine Cervical Disease; Mass Screening
Keywords: HPV self-sampling, cervical cancer screening in older women
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Uterine Cervical Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Eligible women residing in the Central Denmark Region will be assigned to intervention group. Women in the intervention group receive an invitation for HPV-based cervical cancer screening by attending either 1) GP-based screening or 2) HPV self-sampling. The self-sampling kit includes the dry Evalyn brush self-sampling device (Rovers Medical Devices B.V, Oss, Netherlands), written and picture-based user instructions on how to collect and mail the self-sample, and a prestamped return envelope addressed to the Department of Pathology, Randers Regional Hospital.
  Interventions: Other: GP-based screening or HPV self-sampling
- Control group: Eligible women residing in the other five Danish regions (North, Central, South, Zealand and Capital ) will be assigned to control group. Women in the control group will receive usual care, which for 65-69 year-old women is opportunistic cervical cancer screening at the GP

INTERVENTIONS:
Other: GP-based screening or HPV self-sampling — Women in the intervention group will receive an invitation for HPV-based cervical cancer screening by either 1) scheduling an appointment for a cervical cytology by the GP or 2) collect a cervico-vaginal sample themselves in their own home using a self-sampling kit.
  Other Names: Opportunistics GP-based screening
  Groups: Intervention group

SUMMARY:
This study evaluates the effect and feasibility of expanding the target population in the Danish cervical cancer screening program to include women aged 65 to 69 years. The study also evaluates if HPV self-sampling constitutes an appropriate screening method among older women.

DETAILED DESCRIPTION:
The study is a nationwide population-based prospective cohort study embedded in the routine cervical cancer screening program in the Central Denmark Region. The study includes all 65 to 69 years old Danish women with no record of a cervical cytology sample or screening invitation within the last five years. Furthermore, the women are not registered as ineligible for screening, eg due hysterectomy. Eligible women residing in the Central Denmark Region are allocated to the intervention group (n=20,000), while women residing in the other four Danish regions are allocated to the control group receiving standard care (n=71,500), which for this group is low-level opportunistic screening at the general practitioner (GP). The intervention group are invited for HPV-based screening by the GP or to request a self-sampling kit.

ELIGIBILITY:
Inclusion Criteria:

* 65 to 69 years;
* Resident in Denmark
* No record of a cervical cytology or screening invitation in the past 5 years
* Not registered as ineligible for screening

Exclusion Criteria:

* Death
* Migration to or from Denmark
* Moving to or from the CDR
* Residing in the CDR, but having GP in another region
* A record of hysterectomy

Ages: 65 Years to 69 Years | Sex: Female
Age Groups: Older Adult
Gender Based: Yes — Only women are offered cervical cancer screening
Study Population: The study population will include women who had their last cervical cytology sample or screening invitation recorded 5 years or more ago
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Participation rate in the intervention group: | 1 year post invitation
  Participation rate, eg the roportion of targeted women participating by GP-based screening or self-sampling
HPV prevalence | 1 year post invitation
  Number of women tested positive for HPV
Compliance to follow-up among HPV-positive self-samplers | 90 days post test results
  The proportion of HPV-positive self-samplers who attend appropriate follow-up by their GP for onward referral
Screening history | Average of 10 years
  Screening history of participants and non-participants in the intervention group
Intervention versus control group: | 1 year post invitation
  Participation rate
Cytological findings | 1 year post invitation
  Proportion of abnormal cytological findings between the intervention and control group is compared
Histological findings | 1 year post invitation
  Proportion of abnormal histological findings between the intervention and control group is compared
Incidence | 5 year post invitation
  The incidence rate of cervical cancer developed within 5 year is compared between the intervention and control group
Mortality | 5 year post invitation
  The mortality rate of cervical cancer developed within 5 year is compared between the intervention and control group

CONTACTS AND LOCATIONS:
Overall Officials: Mette T Tranberg, post doc phd, Principal Investigator — Randers Regional Hospital, Central Denmark Region
Locations (1):
- Mette Tranberg Nielsen, Randers, Randers NØ, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tranberg M, Petersen LK, Hammer A, Elfstrom M, Blaakaer J, Jorgensen SF, Bennetsen MH, Jensen JS, Andersen B. Value of a catch-up HPV test in women aged 65 and above: A Danish population-based nonrandomized intervention study. PLoS Med. 2023 Jul 6;20(7):e1004253. doi: 10.1371/journal.pmed.1004253. eCollection 2023 Jul. PMID 37410699
- [Derived] Tranberg M, Petersen LK, Elfstrom KM, Hammer A, Blaakaer J, Bennetsen MH, Jensen JS, Andersen B. Expanding the upper age limit for cervical cancer screening: a protocol for a nationwide non-randomised intervention study. BMJ Open. 2020 Nov 5;10(11):e039636. doi: 10.1136/bmjopen-2020-039636. PMID 33154056
- [Derived] Hammer A, Gustafson LW, Christensen PN, Brondum R, Andersen B, Andersen RH, Tranberg M. Implementation of p16/Ki67 dual stain cytology in a Danish routine screening laboratory: Importance of adequate training and experience. Cancer Med. 2020 Nov;9(21):8235-8242. doi: 10.1002/cam4.3399. Epub 2020 Sep 7. PMID 32894896